CLINICAL TRIAL: NCT02708303
Title: Mayo Clinic Foregut Surgery Report Card Questionnaire
Status: Terminated | Type: Observational
Why Stopped: Study's original Principal Investigator no longer at the institution.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Janani S. Reisenauer, Principal Investigator, Mayo Clinic
Other Study IDs: 16-001151
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Gastroesophageal Reflux; Fundoplication; Hernia, Hiatal; Surveys and Questionnaires
Keywords: Esophageal Reflux; Gastric Acid Reflux; Gastric Acid Reflux Disease; Gastro-Esophageal Reflux; Gastro-oesophageal Reflux; Gastroesophageal Reflux Disease; Reflux, Gastroesophageal; Esophageal Hernia; Hernia, Esophageal; Hernia, Paraesophageal; Hiatal Hernia; Sliding Hiatal Hernia; Sliding Esophageal Hernia; Hernia, Hiatus; Paraesophageal Hiatal Hernia; Questionnaires
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Foregut Surgery: Foregut surgery includes conditions of the esophagus, stomach and proximal small intestine. More specifically foregut surgery includes surgery for gastroesophageal reflux disease, hiatal hernias, and paraesophageal hernias.
  Interventions: Other: Mayo Clinic Foregut Surgery Report Card Questionnaire

INTERVENTIONS:
Other: Mayo Clinic Foregut Surgery Report Card Questionnaire — Patients will be asked to complete the Mayo Clinic Foregut Surgery Report Card Questionnaire at approximately 8-10 weeks following surgery and then with each surveillance clinic visit or a minimum of once per year for their lifetime. The questionnaire can be completed at their clinic visit, over the telephone, or by mail. The patient's medical record will also be reviewed to gather any other contributing information.
  Data collected from the questionnaire will be entered into a database that will be maintained for future research.

SUMMARY:
The Mayo Clinic Foregut Surgery Report Card Questionnaire has been created in order to have a consistent evaluation tool for patients undergoing foregut surgery in order to standardize and validate outcome measures.

DETAILED DESCRIPTION:
Foregut surgery includes conditions of the esophagus, stomach and proximal small intestine. More specifically foregut surgery includes surgery for gastroesophageal reflux disease, hiatal hernias, and paraesophageal hernias. Patients undergoing foregut surgery report having varying degrees of symptoms of reflux, regurgitation, dysphagia, and pain following surgery. Providers also note varying degrees of outcomes. Some of these issues can be assessed using pH probe testing, upper GI endoscopy, high resolution manometry, CT scans, and other testing. There are various validated questionnaires that have been used to assess problem areas of reflux, dysphagia, and pain such as the Promis Global Health Score, Mayo GER Score, Modified Dysphagia Questionnaire-30 Day, Zubrod Score, and pain scale. Each of these symptoms, tests, and questionnaires contributes to the provider's understanding of the patient's outcomes but there is currently no assessment tool that brings all of the test findings and information reported by the patient as symptoms or answers to the questionnaires in a format that that is usable for the clinician and understandable for the patient who has specifically undergone foregut surgery. The Mayo Clinic Foregut Surgery Report Card Questionnaire has been created in order to have a consistent evaluation tool for patients undergoing surgery in the foregut in order to standardize and validate outcome measures. Data will be used to establish the validation of the Mayo Clinic Foregut Surgery Report Card Questionnaire. Data will also lead to the establishment of "normal" or expected scores for patients undergoing each type of foregut procedure.

ELIGIBILITY:
* ≥ 18 years old
* Scheduled to undergo Foregut surgery at Mayo Clinic Rochester which includes surgery for gastroesophageal reflux disease, hiatal hernias, and paraesophageal hernias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing or having already undergone foregut surgery at Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Completion of the Mayo Clinic Foregut Surgery Report Card Questionnaires by patients at varying time points following surgery | 1 year
  Completed Mayo Clinic Foregut Surgery Report Card Questionnaires will be analyzed and used to establish validation.

SECONDARY OUTCOMES:
Establishment of "normal" or expected scores from the Mayo Clinic Foregut Surgery Report Card Questionnaires | 3 years
  Completed Mayo Clinic Foregut Surgery Report Card Questionnaires will be used in the establishment of "normal" or expected scores for patients undergoing each type of foregut surgery at different time points following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Janani Reisenauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials